CLINICAL TRIAL: NCT00511277
Title: Single-arm, Open-label and Multicenter Phase IV Study: Efficacy and Safety of Quetiapine in Treating Affective Symptoms of Patients With First-episode Psychosis - a Pilot Study
Brief Title: Efficacy and Safety of Quetiapine in Treating Affective Symptoms of Patients With First-episode psychosis-a Pilot Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Institut fuer anwendungsorientierte Forschung und klinische Studien GmbH (Other)
Collaborators: University of Göttingen (Other)
Responsible Party: Prof. Peter Falkai, MD PhD, University Hospital of Göttingen
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D1449L00016
Record Dates: First submitted 2007-08-02; First posted 2007-08-03 (Estimated); Last update posted 2011-06-21 (Estimated); Status verified 2011-06

CONDITIONS: Schizophrenia
Keywords: quetiapine; schizophrenia; first-episode psychosis; depression; psychopathology
MeSH Terms: conditions — Schizophrenia; Depression | interventions — Quetiapine Fumarate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Seroquel® — dosage form: oral, dosage: 300-800mg/d, frequency: twice daily
  Other Names: Quetiapine

SUMMARY:
The purpose of this study is:

To investigate whether a treatment with quetiapine for six months in patients with first-episode psychosis may be effective in treating depressive symptoms.

To investigate whether a treatment with quetiapine for six months in patients with first-episode psychosis may be effective in mania-like symptoms and to evaluate the general efficacy in psychopathology as well as the safety and tolerability of quetiapine.

DETAILED DESCRIPTION:
Affective symptoms, in particular depressive symptoms are prevalent in up to 60% of all patients with schizophrenia. However, it is still uncertain whether depressive symptoms have a prognostic value, having previously been associated with both favorable and poor outcome. In addition, treatment of affective symptoms in patients with schizophrenia is difficult. There is some evidence that atypical antipsychotics such as quetiapine may contribute not only to a reduction in psychotic symptoms but also that these agents may produce an antidepressant effect in schizophrenia and may reduce suicidality. Most of these studies suffer from methodological limitations as the efficacy on affective symptoms has not been the primary target parameter. Concerning the prevalence of affective symptoms in first-episode psychosis knowledge is still poor. This is why we have developed a study design for a pilot-study on 60 patients with first-episode schizophrenia aiming to demonstrate that a treatment with quetiapine over the period of 6 months shows clinical efficacy on affective, particularly depressive symptoms

ELIGIBILITY:
Inclusion Criteria:

All patients who meet the following inclusion criteria are eligible to participate in the study:

* male and female patients with first-episode schizophrenia (based on ICD-10 criteria)
* in- and out-patients
* age between 18 and 45
* verbal IQ 85
* given written informed consent

Exclusion Criteria:

Patients who meet one or more of the following exclusion criteria cannot participate in the study:

* Other Psychiatric disorders not in full remission, concomitant organic mental disorder or mental retardation
* Patients who, in the investigators judgement, pose an imminent risk of suicide or a danger to self or others
* Hamilton Depression Rating Scale<7 points
* Female patients who are pregnant, lactating or at risk of pregnancy
* Female patients who are not using a highly effective method of birth control. A highly effective method of birth control is defined as those which results in a low failure rate (i.e. less than 1% per year) when used consistently and correctly such as implantants, injectables, combined oral contraceptives, some IUDs, sexual abstinence or vasectomised partner. For subjects using a hormonal contraceptive method, information regarding the product under investigation and its potential effect on the contraception must be addressed.
* history of idiopathic orthostatic hypotension, or condition that would predispose to (dehydration, hypovolaemia)
* Risk of transmitting human immunodeficiency virus (HIV) or hepatitis B and C, via blood or other body fluids
* history of non-compliance as judged by the investigator
* Patients with substance dependence. A urine drug screen will be performed. The investigator will evaluate the results along with medical history to determine if the patient meets the DSM-IV criteria for substance dependence
* Patients with known diabetes mellitus or impaired glucose tolerance, especially a patient with Diabetes Mellitus (DM) fulfilling one of the following criteria:

  * unstable DM defined as enrollment glycosylated hemoglobin (HbA1c)>8.5%
  * patients admitted to hospital for treatment of DM or DM related illness in past 12 weeks
  * patients not under physicians care for DM
  * physicians responsible for patient´s DM care has not indicated that patient´s DM is controlled
  * physician responsible for patient´s DM care has not approved patient´s participation in the study
  * patient has not been on the same dose of oral hypoglycemic drug(s) and/or diet for the 4 weeks prior to randomization. (For thiazolidinediones (glitazones) this period should not be less than 8 weeks)
  * patients taking insulin whose daily dose on one occasion in the past 4 weeks has been more than 10% above or below their mean dose in the preceding 4 weeks.

Note: If a diabetic patient meets one of these criteria, the patient is to be excluded even if the treating physician believes that the patient is stable and can participate in the study.

* ECG considered to show clinical significant abnormalities at enrolment as determined by a cardiologist
* Use of drugs that induce or inhibit the hepatic metabolizing cytochrome 3A4 enzyme within 2 weeks prior to randomization (e.g. inducers: phenytoin, carbamazepine, phenobarbital, rifampicin, rifabutin, glucocorticoids, thioridazine and St. Johns´wort (=Johanniskraut) and inhibitors: ketaconazole (except for topical use), itraconazole, fluconazole, erythromycin, clarithromycin, fluvoxamine, nefazodone, troleandomycin, indinavir, nelfinavir and saquinavir).
* patients with insufficient knowledge of the German language
* A thyroid-stimulating hormone (TSH) concentration more than 10% above the upper limit of the normal range and the laboratory used for sample analysis at enrolment, whether or not the subject is being treated for hypothyroidism
* Any serious and unstable somatic illness (e.g. malignant tumor, severe cardiovascular disease, etc.) that, in the opinion of the investigator, would be negatively affected by the study medication or that would affect study medication. If relevant medical findings are obtained during the examination, it is at the physician's discretion to initiate additional examinations (e.g. lab testing, ECG). If medically indicated examinations have already been carried out, the results should not be older than two weeks at the time of the screening visit. The patient can only participate in the study if all study results are within the normal range or the examiner has determined a deviation as clinically irrelevant. This should be clearly documented in the CRF.
* Participation in another drug trial within 4 weeks prior to enrolment into this study or longer in accordance with local requirements

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2007-08; Primary Completion 2010-10 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Changes in the Hamilton Depression Rating Scale (HAMDS) from Baseline to Endpoint | treatment for six months

SECONDARY OUTCOMES:
Changes in the Young Mania Rating Scale,Changes in the Positive and Negative Syndrome Scale,Changes in the Clinical Global Impression Scale(CGI,Changes in the self assessment of depressive symptoms(Beck Depression Inventory) from Baseline to Endpoint. | for six months

CONTACTS AND LOCATIONS:
Overall Officials: Peter Falkai, MD PhD, Study Director — Department of Psychiatry and Psychotherapy, GEORG-AUGUST-UNIVERSITY GÖTTINGEN, GERMANY; Thomas Wobrock, MD PhD, Principal Investigator — Department of Psychiatry and Psychotherapy, GEORG-AUGUST-UNIVERSITY GÖTTINGEN, GERMANY; Andreas Heinz, MD PhD, Principal Investigator — Department of Psychiatry and Psychotherapy, Charité Campus Mitte Berlin, Germany; Georg Juckel, MD PhD, Principal Investigator — Department of Psychiatry, Ruhr University Bochum, Germany
Locations (1):
- Department of Psychiatry and Psychotherapy, GEORG-AUGUST-UNIVERSITY GÖTTINGEN, Göttingen, Germany